CLINICAL TRIAL: NCT00099281
Title: A Phase III Study of DPPE Combined With Epirubicin and Cyclophosphamide vs Epirubicin and Cyclophosphamide Alone as First Line Treatment in Metastatic/Recurrent Breast Cancer
Brief Title: DPPE in Combination With Epirubicin and Cyclophosphamide in the Treatment of Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: YM BioSciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMB1002 02
Record Dates: First submitted 2004-12-10; First posted 2004-12-10 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Breast Cancer; Metastases
Keywords: Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Drug: YMB 1002

SUMMARY:
The purpose of this trial is to study DPPE combined with epirubicin and cyclophosphamide in patients with metastatic and/or recurrent breast cancer who may have received previous hormone treatment but have not had exposure to anthracycline treatment. Stratification allocation will be within the following subgroups:

1. Prior cytotoxic treatment;
2. Estrogen receptor status;
3. ECOG performance status;
4. Number of cycles of chemotherapy.

DETAILED DESCRIPTION:
Endpoints of the trial are as follows:

primary: overall survival; secondary: response rate, progression free survival, toxicity, neurocognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of breast cancer
* Documented evidence of metastatic and/or recurrent breast cancer
* Presence of at least one bi-dimensional or uni-dimensional lesion
* ECOG status 0, 1 or 2
* Quality of life

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700
Dates: Start 2004-05; Study Completion 2006-06

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Response rate
Progression-free survival
Toxicity
Neurocognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Pritchard, MD, Study Chair — Sunnybrook Health Sciences Centre
Locations (1):
- PharmOlam, London, United Kingdom